CLINICAL TRIAL: NCT06635187
Title: An Investigation Into the Oral-motor and Speech Functions of Post-stroke Individuals Via an AI-powered Mobile Health Application
Brief Title: ORal-motor Assessment and Rehabilitation Mobile App (ORAR App)
Acronym: ORAR
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: P0046834; FBL/036/23 (Other Grant/Funding Number: Innovation and Technology Commission)
Record Dates: First submitted 2024-09-27; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Oral Motor Functions
Keywords: Mobile App; Stroke; Oral Motor functions; Rehabilitation; artificial intelligence; speech
MeSH Terms: conditions — Stroke; Speech

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stroke patients: Adult stroke patients will be recruited to undergo a series of examinations on oral-motor and speech functions.
  Interventions: Diagnostic Test: Speech and swallowing assessment
- Control group: Neurologically healthy adults residing in Hong Kong will undergo the same set of assessments and procedures as the stroke patient group.
  Interventions: Diagnostic Test: Speech and swallowing assessment

INTERVENTIONS:
Diagnostic Test: Speech and swallowing assessment — This is an observational study in which post-stroke patients will undergo a series of assessments tapping oral-motor and speech functions. Both behavioral and instrumental examinations will be used. Their performance will be captured via an artificial intelligence(AI)-powered mobile health application. The relation between the oral/speech-motor movements captured by the app and their performance as measured via instruments/behavioral means will be investigated.

SUMMARY:
The goal of this study is to set up a database of oral-motor and speech functions of post-stroke patients in Hong Kong via an artificial intelligence-powered mobile-health application. The main study objectives are:

1. To establish an image database of oral-facial movements of neurologically healthy adults and adult stroke patients in Hong Kong.
2. To evaluate the oral-motor functions of neurologically healthy adults and stroke patients via instrumental and behavioral assessment.
3. To investigate the correlation between image-based analysis of oral-facial functions and instrumental evaluations and subjective judgment by the speech-language therapist.

ELIGIBILITY:
For Neurologically healthy adults,

Inclusion Criteria:

1. age between 20 and 85 years old;
2. no severe systemic diseases such as uncontrolled diabetes, cerebrovascular diseases, head and neck tumors, or neurological disorders;
3. not undergoing radiation therapy or chemotherapy;
4. normal or corrected-to-normal vision and hearing; and
5. fluent Cantonese speakers

Exclusion Criteria:

1) participants who are unable to sign the "Informed Consent Form" due to cognitive impairments

For stroke patients,

Inclusion Criteria:

1. age between 20 and 85 years old;
2. a history of stroke;
3. not undergoing radiation therapy or chemotherapy;
4. normal or corrected-to-normal vision and hearing;
5. premorbid fluent Cantonese speakers; and
6. able to follow simple commands.

Exclusion Criteria:

1. individuals currently on non-oral feeding; and
2. participants who are unable to sign the "Informed Consent Form" due to cognitive impairments

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medically stable stroke patients and neurologically health adults aged between 20-85 years will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Diadochokinetic (DDK) rate of alternating and sequential labial, alveolar and velar plosive sounds | 2-hr assessment
  Participants will be asked to produce /pa/, /ta/, and /ka/ as quick as possible in 10 seconds as alternating motion rate and /pataka/ in 10 seconds as sequential motion rate.
Tongue strength endurance measured by tongue pressure sensor (model: TPM-02, JMS, Hiroshima, Japan) | 2-hr assessment
  Tongue endurance is defined as the time it takes to reach 60 % or more of maximum tongue strength. Three trials were performed, while the average duration (in terms of seconds) taken by the tongue pressure sensor will be used to determine tongue function.
Mastication efficiency as measured via glucose sensor (model: GS-II, GC Corporation, Toyko, Japan) | 2-hr assessment
  A 2-gram gummy jelly that comes with the glucose sensor will be put into the mouth, and the subject will be asked to chew the gummy for 20 seconds. Afterward, everything will be discharged into a paper cup, and the resultant filtrate will be examined quantitatively via the glucose sensor. Mastication efficiency will be illustrated in terms of milliliter per deciliter (mL/dL).
Occlusal force as measured via the occulsal pressure measurement film (model: Dental Prescale II, GC Corporation, Toyko, Japan) | 2-hr assessment
  An occlusal pressure measurement film will be put into the oral cavity and s/he will be asked to close the jaw firmly for 2-3 seconds. The film will be scanned by a scanner (model: GT-X830, Epson, Nagano, Japan) and analyzed by a software called Bite force analyzer manufactured by the GC Corporation. Occlusal force will be represented in Newton.
Maximum tongue strength measured by tongue pressure sensor (model: TPM-02, JMS, Hiroshima, Japan) | 2-hr assessment
  Participants will be asked to press the bulb of the tongue pressure sensor with the anterior part of the tongue as hard as they can. The maximum tongue strength in kilopascal (KPa) will be measured by the sensor.

SECONDARY OUTCOMES:
The Chinese version of the Oral Health Impact Profile-14 (OHIP-14) questionnaire to assess oral health-related quality of life. | 2-hr assessment
  Participants will be asked to give ratings on the questionnaire based on a 5-point Likert scale. Lower scores represent better oral condition-related quality of life. The maximum and minimum scores are 56 and 0, respectively.
Chinese version of Eating Assessment Tool (EAT-10) questionnaire as a self-reported outcome instrument on swallowing functions | 2-hr assessment
  The questionnaire consists of 10 questions, and participants will be asked to evaluate their swallowing functions based on a 5-point Likert scale (0=not at all; 4=very much). Lower scores reflect better swallowing performance. Maximum and minimal scores are 40 and 0, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Winsy Wing Sze Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Speech Therapy Unit, Room 701, Block EF, The Hong Kong Polytechnic Unviersity, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be available on an open-access repository such as OSF.
Supporting Information: Study Protocol, ICF
Time Frame: 5 years upon the project end date
Access Criteria: Open access to all people